CLINICAL TRIAL: NCT01136629
Title: Clinical, Histological and Biochemical Characterization of Hyperpigmented Lesion.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: LIM THIAM CHYE / Professor, National University Hospital, Singapore
Other Study IDs: NUHS/SUR-PRAS/2010/4; D / 08 / 175 (Registry Identifier: DSRB - D / 08 / 175)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Lentigo; Melasma
Keywords: Hyper-pigmented spots; Lentigines; Mealsma; RNA extraction; Isolation of Keratinocytes; Isolation of Melanocytes
MeSH Terms: conditions — Lentigo; Melanosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subjects with hyper-pigmented spots: Subjects age 21 to 80 year old, who have elected to undergo a plastic surgery will be enrolled. Subjects will be from Chinese, Malay, Indian or Caucasian ancestry. Subjects will be female or male with a hyper-pigmented spots.

SUMMARY:
Hypothesis -

The developments of solar lentigine and melasma are due to mutations in keratinocytes that drive the production and transfer of pigment from melanocytes to keratinocytes.

DETAILED DESCRIPTION:
Aims -

1. Characterize and classify lentigines and mealsma from a clinical and physiological point of view. This will help us to better understand the cellular processes leading to the development of lentigines (also referred to as Senile or Solar Lentigo).
2. Proper characterization and classification of lentigines and melasma would facilitate the development of models to study and find solutions to treat these lesions.

Hypothesis - The developments of solar lentigine and melasma are due to mutations in keratinocytes that drive the production and transfer of pigment from melanocytes to keratinocytes.

Methodology -

Patients, 21 - 80 year old, who have elected to undergo a plastic surgery will be enrolled. Some patient information (i.e. age, sex, race, family history, life-style related to sun-exposure) will be collected.

After surgery, hyper-pigmented spots will be excised and stored in individual containers for subsequent experimental procedures.

Before surgery, the area containing the hyper-pigmented spots will be photographed using a high resolution digital camera and assessed using optical probes (Spectrophotometer to measure skin chromophores, mexameter to measure the melanin and erythema indexes and a diffuse reflectance spectrometer to measure hemoglobin, deoxyhemoglobin and melanin).

After surgery, excised skin samples will be processed for histological assessments, others for gene or protein expression analysis, and yet another group will be used to isolate keratinocyte and melanocyte to further study their behavior and response to stimuli in primary cultures.

Clinical assessment of Hyperpigmented lesions:

Lentigo Morphological assessment (before surgery)

1. Macules vary in color from yellow, light-brown to black, depending on under-lying skin type
2. Size varies from 1mm to greater than 1 cm
3. Appear on sun-exposed areas (face, neck, etc)

Morphological assessment (before surgery)

1. Irregular light to dark brown to gray brown macules or patches on sun-exposed areas
2. When examine with Wood's lamp, melasma can be classified into 3 types, epidermal, dermal, or mixed, based on intensity of pigments, in which epidermal melasma has darker color than derma melasma. Mixed melasma has a mixture of both dark and light pigmentations
3. Melanocytes in melasma lesion have an increase in the number of mitochondria, golgi apparatus, rough ER, and ribosomes

Spectrophotometer will be used to measure the optical properties of spots and control areas (without the spot)

Sample processing

1. RNA extraction
2. Histology
3. Isolation of Keratinocytes, and Melanocytes.

ELIGIBILITY:
Inclusion Criteria:

* Solar Lentigines and/or Melasma on facial, or neck areas
* Ethnic background: Chinese, Malay, Indian, Caucasian
* Age 21 - 80 years old
* Ability to provide informed consent

Exclusion Criteria:

* Pregnant and lactating women
* Children under the age of 20
* Neoplasm (past or present) in excised area
* Patients with communicable disease
* Immuno-compromised patients
* Current treatment with an investigational drug

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects age 21 to 80 year old, who have elected to undergo a plastic surgery will be enrolled. Patients will be from Chinese, Malay, Indian or Caucasian ancestry. Patients will be female or male with hyper-pigmented spots.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2008-06; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Characterization and classification of lentigines and melasma | 3 years
  Characterize and classify lentigines and mealsma from a clinical and physiological point of view. This will better understand the cellular processes leading to the development of lentigines (also referred to as Senile or Solar Lentigo).
  Proper characterization and classification of lentigines and melasma would facilitate the development of models to study and find solutions to treat these lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Thiam Chye Lim, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore, Singapore